CLINICAL TRIAL: NCT01941524
Title: Assessment of the Cerebral Tissue Oxygenation and the Bioelectrical Brain Activity of Preterm Newborns During Administration of Two Different Surfactant
Brief Title: Brain Oxygenation and Function of Preterm Newborns During Administration of Two Different Surfactant Preparations
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Poznan University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Tomasz Szczapa, doctor of medical science, Poznan University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 502-14-02215338-09873
Record Dates: First submitted 2013-06-19; First posted 2013-09-13 (Estimated); Last update posted 2020-03-05 (Actual); Status verified 2020-03

CONDITIONS: Respiratory Distress Syndrome, Newborn; Respiratory Failure
Keywords: Brain oxygenation; NIRS; aEEG; surfactant
MeSH Terms: conditions — Respiratory Distress Syndrome, Newborn; Respiratory Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Poractant goup (Active Comparator): Newborns, who will be monitored by amplitude integrated electroencephalography (aEEG) and near infrared spectroscopy (NIRS) during poractant instillation.
  Interventions: Drug: Poractant alfa instillation
- Beractant group (Active Comparator): Newborns who will be monitored by aEEG and NIRS during beractant instillation
  Interventions: Drug: Beractant instillation

INTERVENTIONS:
Drug: Poractant alfa instillation — aEEG and NIRS monitoring during poractant alfa instilation
  Arms: Poractant goup
Drug: Beractant instillation — aEEG and NRs monitoring during beractant instillation
  Arms: Beractant group

SUMMARY:
The purpose of the study is to determine whether there are differences in bioelectrical function (measured by amplitude integrated electroencephalography) and brain oxygenation (measured by near infrared spectroscopy) while and after instillation of two different surfactant preparations.

DETAILED DESCRIPTION:
Patients randomized to one of the treatment groups: 1) SRT with porcine preparation - poractant alfa; 2) SRT with bovine preparation - beractant. Continuous monitoring and simultaneous recordeding of 1) saturation (SpO2) and heart rate (HR) measured with pulse oximetry, cerebral tissue oxygenation measured with near-infrared spectroscopy, amplitude-integrated electroencephalography.

ELIGIBILITY:
Inclusion Criteria:

* 26-30 gestational age
* surfactant instillation

Exclusion Criteria:

* congenital heart disease
* congenital central nervous disorder
* congenital genetic disorders

Ages: 15 Minutes to 2 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2013-03-03; Primary Completion 2015-06-20 (Actual); Study Completion 2015-06-20 (Actual)

PRIMARY OUTCOMES:
Cerebral oxygenation | 4 hours after surfactant instillation
  Cerebral tissue oxygenation measured with near-infrared spectroscopy
Brain bioelectrical activity | 4 hours after surfactant instillation
  Brain bioelectrical activity measured with amplitude-integrated electroencephalography (aEEG)

CONTACTS AND LOCATIONS:
Overall Officials: Tomasz Szczapa, M.D., Study Director — Poznan University of Medical Sciences
Locations (1):
- Department of Neonatology, Poznan, Great Poland, Poland